CLINICAL TRIAL: NCT00519779
Title: Academic Stress and Proinflammatory Cytokines: Omega-3 Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Principal Investigator, Janice Kiecolt-Glaser, Professor, National Center for Complementary and Integrative Health (NCCIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21AT003912-01A1 (NIH); AT003912
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Results first posted 2012-03-22 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-02

CONDITIONS: Stress-related Changes in Inflammation
Keywords: affect; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Placebo oral Omega-3 fish oil supplementation
  Interventions: Dietary Supplement: Oral omega-3 fish oil placebo
- 1 (Experimental): oral Omega-3 fish oil supplementation
  Interventions: Dietary Supplement: omega-3 supplementation

INTERVENTIONS:
Dietary Supplement: omega-3 supplementation — 2.5 g/day omega-3
  Arms: 1
Dietary Supplement: Oral omega-3 fish oil placebo — to match experimental dosage
  Arms: 2

SUMMARY:
This study is designed to examine the effects of fish oil on immune function and mood in medical students.

DETAILED DESCRIPTION:
This study will examine how supplementation with omega-3 polyunsaturated fatty acids (key fish oil components) affects immune and mood responses to examination stress. This study will examine these outcomes in medical students during academic examination periods as well as less stressful non-exam periods. Participants will take fish oil supplements or placebo pills for approximately 3 months during which time relevant mood, endocrine, and immune measures will be assessed.

For detailed information about the study, please visit our website at http://www.stressandhealth.org

ELIGIBILITY:
Inclusion Criteria:

* OSU preclinical medical or dental student, or graduate nursing student
* male or female

Exclusion Criteria:

* taking certain medications with immune or endocrine effects
* chronic health conditions
* smoking
* excessive use of alcohol or caffeine
* significant digestive problems
* routine use of fish oil or flaxseed supplements or high fish intake
* fish allergy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice K Kiecolt-Glaser, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Medicine, Columbus, Ohio, United States

REFERENCES:
- [Result] Kiecolt-Glaser JK, Belury MA, Andridge R, Malarkey WB, Glaser R. Omega-3 supplementation lowers inflammation and anxiety in medical students: a randomized controlled trial. Brain Behav Immun. 2011 Nov;25(8):1725-34. doi: 10.1016/j.bbi.2011.07.229. Epub 2011 Jul 19. PMID 21784145
- See also: Please click here to visit our website if you would like to read more about the study or apply to participate. — http://www.stressandhealth.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo oral Omega-3 fish oil supplementation
- Omega-3 Fish Oil Supplement: oral Omega-3 fish oil supplementation, 2.496 grams of omega-3/day (2085 mg of eicosapentaenoic acid [EPA] and 348 mg of docosahexaenoic acid [DHA])
Period: Overall Study
Arm/Group | Placebo | Omega-3 Fish Oil Supplement
Started | 34 | 34
Completed | 34 | 33
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Omega-3 Fish Oil Supplement | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 34 | 68
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 23.4 (1.7) | 23.9 (2.0) | 23.6 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 20 | 18 | 38
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Serum ln(IL-6)
Description: log-transformed serum Interleukin-6 (IL-6)
  Serum cytokine levels provide an assessment of systemic inflammation, the cytokine level circulating throughout the body. Higher levels are typically interrupted as worse unless an individual is acutely ill.
  Stimulated cytokine production reflects the inflammatory cytokine production capacity of monocytes.
Time Frame: every 3 weeks for 3 months after initiating supplementation (outcome reported is the average outcome across all 4 time points)
Population: intention to treat
Measure: Least Squares Mean (Standard Error); unit: ln(pg/mL)
Arm/Group | Placebo | Omega-3 Fish Oil Supplement
Number analyzed (Participants) | 34 | 34
ln(pg/mL) | 0.054 (0.070) | 0.051 (0.069)
Statistical Analysis 1: Comparison: Placebo vs Omega-3 Fish Oil Supplement; Test type: Superiority or Other; p = 0.97, Mixed Models Analysis; adjusted for baseline value, visit, gender, SAD; Mean Difference (Final Values) = -0.0033, 95% CI 2-sided [-0.18 to 0.18], Standard Error of Mean 0.090

2. Secondary Outcome: ln(Beck Anxiety Score)
Description: log-transformed Beck anxiety score, min-max values - 0-4.1: higher means greater anxiety
Time Frame: as for outcome 1
Population: intention to treat
Measure: Least Squares Mean (Standard Error); unit: units
Arm/Group | Placebo | Omega-3 Fish Oil Supplement
Number analyzed (Participants) | 34 | 34
units | 1.2 (0.075) | 0.93 (0.076)
Statistical Analysis 1: Comparison: Placebo vs Omega-3 Fish Oil Supplement; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.44 to -0.011], Standard Error of Mean 0.11

3. Primary Outcome: Serum ln(TNF-a)
Description: log-transformed serum Tumor Necrosis Factor-alpha (TNF-alpha)
  All cytokine measurements (e.g., IL-6 and TNF-a, serum and stimulated) were analyzed across time; however, no stress effects were found. Therefore, all assessments post-supplementation were averaged (time points 3-6) and analyzed to determine whether fish oil supplementation had an effect. Pooling these 4 assessments provides a better estimate of an individual's cytokine levels because single time point measurements can be affected by changes in exercise, alcohol consumption, or sleep in the preceding 24-48 hours.
Time Frame: as for outcome 1
Population: intention to treat
Measure: Least Squares Mean (Standard Error); unit: ln(pg/mL)
Arm/Group | Placebo | Omega-3 Fish Oil Supplement
Number analyzed (Participants) | 34 | 34
ln(pg/mL) | 0.61 (0.028) | 0.54 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Omega-3 Fish Oil Supplement; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = -0.076, 95% CI 2-sided [-0.15 to 0.002], Standard Error of Mean 0.039

4. Primary Outcome: Stimulated ln(IL-6)
Description: log-transformed stimulated IL-6
  Serum cytokine levels provide an assessment of systemic inflammation, the cytokine level circulating throughout the body. Higher levels are typically interrupted as worse unless an individual is acutely ill.
  Stimulated cytokine production reflects the inflammatory cytokine production capacity of monocytes.
Time Frame: as for outcome 1
Population: intent to treat
Measure: Least Squares Mean (Standard Error); unit: ln(pg/mL)
Arm/Group | Placebo | Omega-3 Fish Oil Supplement
Number analyzed (Participants) | 34 | 34
ln(pg/mL) | 11.1 (0.051) | 10.9 (0.050)
Statistical Analysis 1: Comparison: Placebo vs Omega-3 Fish Oil Supplement; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.30 to -0.009], Standard Error of Mean 0.072

5. Primary Outcome: Stimulated ln(TNF-alpha)
Description: log-transformed stimulated TNF-alpha
Time Frame: as for outcome 1
Population: intention to treat
Measure: Least Squares Mean (Standard Error); unit: ln(pg/mL)
Arm/Group | Placebo | Omega-3 Fish Oil Supplement
Number analyzed (Participants) | 34 | 34
ln(pg/mL) | 7.4 (0.061) | 7.3 (0.060)
Statistical Analysis 1: Comparison: Placebo vs Omega-3 Fish Oil Supplement; Test type: Superiority or Other; p = 0.08, Mixed Models Analysis; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.33 to 0.018], Standard Error of Mean 0.086

6. Secondary Outcome: ln(CES-D)
Description: log-transformed Center for Epidemiologic Studies Depression Scale (CES-D) score
  The CES-D is a self-report scale designed to measure current symptoms of depression rated on a four-point likert scale.
  Scores range from 0-60, with higher scores indicating a higher frequency of depressive symptoms.
Time Frame: as for outcome 1
Population: intention to treat
Measure: Least Squares Mean (Standard Error); unit: scores on a
Arm/Group | Placebo | Omega-3 Fish Oil Supplement
Number analyzed (Participants) | 34 | 34
scores on a | 1.6 (0.097) | 1.6 (0.098)
Statistical Analysis 1: Comparison: Placebo vs Omega-3 Fish Oil Supplement; Test type: Superiority or Other; p = 0.93, Mixed Models Analysis; Mean Difference (Final Values) = 0.012, 95% CI 2-sided [-0.26 to 0.29], Standard Error of Mean 0.14

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Placebo | Omega-3 Fish Oil Supplement
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 18/34 | 20/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=34) | Omega-3 Fish Oil Supplement (N=34)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (8)
Nasal symptoms (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7)
Stomach pain (Gastrointestinal disorders) | 5 (5) | 6 (6)
Tachycardia (Cardiac disorders) | 6 (6) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Skin rash (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Heartburn (Cardiac disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No